CLINICAL TRIAL: NCT06002659
Title: A Phase I/IIa Multicenter Study Evaluating the Safety and Efficacy of CAR20(NAP)-T in Patients With Relapsed/Refractory B Cell Lymphoma (CARMA-01 Study)
Brief Title: CAR20(NAP)-T Therapy for B Cell Lymphoma (CARMA-01 Study)
Acronym: CARMA-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Elicera Therapeutics (Unknown); Uppsala University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELC301-CARMA-01; 2022-004157-31 (EudraCT Number)
Record Dates: First submitted 2023-01-06; First posted 2023-08-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: B-cell Lymphoma
Keywords: CAR T cell; B cell lymphoma; CD20; HP-NAP
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): CAR20(NAP)-T treatment
  Interventions: Biological: CAR20(NAP)-T; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CAR20(NAP)-T — Autologous CAR-T cells targeting CD20 and upon target recognition express and secrete NAP
  Other Names: ELC-301
Drug: Cyclophosphamide — pre-conditioning chemotherapy
Drug: Fludarabine — pre-conditioning chemotherapy

SUMMARY:
The purpose is to study the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of CAR20(NAP)-T for patients with B-cell malignancies.

DETAILED DESCRIPTION:
A cancer patient's T cells can be isolated and engineered to express a chimeric antigen receptor (CAR), which re-directs the T cells to recognize and kill tumor cells expressing that particular antigen. CD19-targeted CAR-T cell therapy has shown good effects for B cell malignancies, even cure, in otherwise therapy refractory patients.

Antigen escape, i.e., the downregulation of the antigen targeted by the CAR due to the selective pressure caused by the CAR-T cell therapy is a challenge. For patients treated with CD19 CAR-T cell therapy, about 30% of the patients are resistant to treatment and about 20% of patients relapse after an initial response.

CAR20(NAP)-T cells target CD20 and upon target recognition secrete a bacterial-derived pluripotent immune-stimulating factor named NAP (Helicobacter pylori Neutrophil-activating protein). Secretion of NAP in the tumor microenvironment can induce an endogenous bystander immune response, that counteracts antigen escape and thereby improves the therapeutic outcome.

CAR20(NAP)-T is an investigational agent not yet approved by authorities.

Design:

The study is designed as 3+3 dose escalation phase I, and a dose expansion Phase IIa. The safety, tolerability, PK/PD, and efficacy will be evaluated.Dose escalation is to be based on the incidence of dose-limiting toxicity (DLTs). The investigator or sub-investigator will decide if the AE is related to IMP-treatment on a case-by-case basis depending on the character of the DLT symptoms. Investigator or sub-investigator has a possibility to classify various toxicity observed in patient as DLT.The Recommended phase II dose (RP2D) is decided based on safety, PK/PD data as well as preliminary clinical activity data from the Phase I dose escalation. After setting the RP2D, additional patients will be treated at RP2D to make sure at least 6 patients will be treated at RP2D dose level already at the phase I part.

Protocol treatment:

The enrolled patient will undergo a leukapheresis procedure to harvest enough T cells for IMP production. During CAR20(NAP)-T manufacturing, the patient may receive bridging therapy to control tumor burden. All patients will receive pre-conditioning chemotherapy (cyclophosphamide and fludarabine) followed by one dose of CAR20(NAP)-T cell infusion intravenously. The patient will then be followed by doctor/study nurse for evaluation of the health status and side effects. At follow-up visits, blood samples will be obtained and CT imaging will be performed. Patient will actively participate in the study for about 24 months when the final follow-up visit will be scheduled.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent.
* Relapsed or refractory CD20+ diffuse large B-cell lymphoma, mantle cell lymphoma or indolent lymphoma.
* The patient should have been treated with at least two lines of therapy and have no curative treatment option, specifically

  * Relapsed or refractory CD20+ B-cell lymphoma that are not eligible to receive clinically approved CD19-directed CAR T cell treatment.
  * Relapsed or refractory CD20+ B-cell lymphoma who are CD19 negative.
  * Relapsed or refractory B-cell lymphoma who relapse after CD19 CAR T cell treatment.
* In phase I age >18 years, in phase II all ages
* Measurable disease per Lugano classification.
* Performance status ECOG 0-2.
* Adequate bone marrow function as evidenced by:

  * Absolute neutrophil count (ANC) ≥ 1x10^9/l/L
  * Platelet ≥ 50x 10^9/l
  * Absolute lymphocyte count ≥ 0,1x10^9/L
* Adequate renal, hepatic, cardiac, and pulmonary function as evidenced by:

  * Creatinine clearance (Cockcroft Gault) ≥ 30 mL/min
  * Serum Alanine aminotransferase/Aspartate aminotransferase (ALT/AST) ≤ 2.5 Upper limit of normal (ULN) and S-Bilirubin <1.5x UNL
  * Cardiac ejection fraction ≥ 40%
* Functional venous for administration of IMP.
* Fertile individuals must consent to use contraceptives during participation in the trial.

Exclusion Criteria:

* Other CD20-positive lymphomas i.e Burkitt lymphoma, primary CNS lymphoma, plasmablastic lymphoma or CLL transformed to DLBCL/HGBL (Richter transformation)
* Any significant medical or psychiatric illness that would prevent the subject from giving informed consent or from following the study procedures.
* Known human immunodeficiency virus (HIV) infection.
* Impending organ-compromising disease.
* Rapidly progressing disease
* Active and/or severe infection (e.g., tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
* Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the subject to perform the treatment.
* Treatment with an investigational product within 30 days prior to enrolment
* Potential sign of hypersensitivity reaction to tocilizumab or any of the agents used in this study
* Systemic corticosteroid treatment (>10mg/day) <5 days prior to IMP treatment or <7 days prior leukapheresis.
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | First infusion up to 30 days
  The incidence of dose limiting toxicity (DLT). Number of Participants Experiencing Adverse Events (AEs) Defined as Dose Limiting Toxicities (DLTs)
Adverse events | 24 months
  The nature, frequency, severity, and tolerability of adverse events (AEs) including clinically significant laboratory data, and their relation to dosage.
Pharmacodynamic (PD) and pharmacokinetic (PK) | Either 24 month or 15 years during long-term follow up if clinically indicated
  PD is assessed by determine circulating B cell level; PK is assessed by determine circulating CAR20(NAP)-T cells.

SECONDARY OUTCOMES:
Objective response rate [ORR] | 24 months
  ORR is defined as the incidence of a complete response or a partial response by the revised Lugano classification as determined by the study investigators. All patients that do not meet the criteria for an objective response by the analysis cutoff date will be considered non-responders.
Progression free survival [PFS] | 24 months
  PFS is defined as the time from the IMP treatment date to the date of disease progression per the revised Lugano classification or death from any cause.
Best Objective Response | 24 months
  the incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as best response to treatment.
Duration of Response (DOR) | 24 months
  DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the revised Lugano classification or death regardless of cause. Patients not meeting the criteria for progression or death by the analysis data cutoff date will be censored at their last evaluable disease assessment date and their response will be noted as ongoing.
Overall Survival (OS) | either 24 months or 15 years during long-term follow up if clinically indicated
  defined as the time from IMP treatment to the date of death. Patients alive by the analysis data cutoff date will be censored at their last contact date. The overall survival rate will be reported at different cut-off time points.

OTHER OUTCOMES:
Anti-NAP response | either 24 months or 15 years during long-term follow up if clinically indicated
  Determine anti-NAP immune response
Bystander immunity activation | either 24 months or 15 years during long-term follow up if clinically indicated
  Assess induced tumor specific endogenous T-cell immune response

CONTACTS AND LOCATIONS:
Overall Officials: Di Yu, PhD, Study Director — Uppsala University
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jin C, Ma J, Ramachandran M, Yu D, Essand M. CAR T cells expressing a bacterial virulence factor trigger potent bystander antitumour responses in solid cancers. Nat Biomed Eng. 2022 Jul;6(7):830-841. doi: 10.1038/s41551-022-00875-5. Epub 2022 Apr 4. PMID 35379957